CLINICAL TRIAL: NCT06152614
Title: MIND Foods and Aerobic Training in Black Adults With HTN: An ADRD Prevention Pilot RCT
Brief Title: MIND Foods and Aerobic Training in Black Adults With HTN
Acronym: MAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Daniel Clark, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16547; R01AG076685 (NIH)
Record Dates: First submitted 2023-11-02; First posted 2023-11-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cognitive Decline; Hypertension; Diet; Aerobic Exercise
Keywords: nutrition; cooking; exercise; hypertension
MeSH Terms: conditions — Cognitive Dysfunction; Hypertension; Motor Activity | interventions — Cooking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (EUC) (Active Comparator): Participants randomized to EUC will have access to existing usual primary care services. They will also be enrolled in Hypertension Self-Management Education and Support (SMES) class ("Hypertension group"), which is an existing CDC-endorsed program offered at Eskenazi Health to provide information and skills for managing hypertension (HTN). Classes are led by registered dietitians via Webex.
  Interventions: Behavioral: Enhanced Usual Care (EUC)
- Food Delivery and Cooking PLUS Aerobic Training (FoRKS+) (Experimental): Participants randomized to FoRKS+ will attend weekly HTN SMES classes separately from EUC participants. SMES classes will include the EUC curriculum stated above and an introduction to the upcoming FoRKS+ intervention.
  Following HTN SMES completion, FoRKS+ continues with home-delivered Mediterranean-style ingredient kits, food management lessons, and hands-on cooking classes in one's own kitchen. Classes are led by registered dietitians via Webex. Classes are held twice per week thru Week 12, then only once per week through Week 16. Intervention continues with aerobic exercise led by health coaches via Webex. Classes start in Week 13 with one session per week, increasing to two sessions per week in Weeks 17-28.
  Interventions: Behavioral: Food Delivery and Cooking PLUS Aerobic Training (FoRKS+)

INTERVENTIONS:
Behavioral: Enhanced Usual Care (EUC) — Enhanced Usual Care (EUC) includes 5 weeks of hypertension classes.
  Arms: Enhanced Usual Care (EUC)
Behavioral: Food Delivery and Cooking PLUS Aerobic Training (FoRKS+) — Food Delivery and Cooking PLUS Aerobic Training (FoRKS+) includes 5 weeks of hypertension classes followed by 11 weeks of home-delivered Mediterranean-style ingredient kits and virtual cooking classes, and an additional 12 weeks of aerobic exercise.
  Arms: Food Delivery and Cooking PLUS Aerobic Training (FoRKS+)

SUMMARY:
The goal of this randomized controlled trial is to determine the impact of Mediterranean-Dash Intervention for Neurodegenerative Delay (MIND) diet and aerobic training on cognition in Black adults with high systolic blood pressure.

Researchers will compare Food Delivery and Cooking PLUS Aerobic Training (FoRKS+) versus Enhanced Usual Care (EUC) to evaluate the effects on cognition.

Participants will complete cognitive and cardiovascular assessments, 24-hr blood pressure monitoring, standard blood pressure measurements, weight, fingerstick for HbA1c point-of-care testing, and questionnaires.

Participants may also choose to participate in an optional blood draw for DNA Repair Capacity testing as a modifiable risk factor for aging-associated diseases.

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate Mediterranean-Dash Intervention for Neurodegenerative Delay (MIND) diet and aerobic training (FoRKS+) versus enhanced usual care (EUC) in Black adults with systolic blood pressure of ≥140 mm Hg. This project seeks to evaluate the potential for high-polyphenol nutritious foods, hands-on training in food management skills, and aerobic exercise to impact cognition and risk factor reduction in persons with prevalent chronic disease.

Adults who pass the telephone screen will be invited to complete a blood pressure check for final eligibility determination. Participants must receive an average systolic read of ≥130 mmHG across 3 standard BP readings with designated wait periods; a maximum of 5 readings may be attempted to receive 3 successful measurements necessary to calculate the average. Participants who meet criteria and give informed consent will complete a full baseline assessment, consisting of cognitive and cardiovascular assessments, blood pressure, weight, HbA1c testing, questionnaires, 24-hour ambulatory blood pressure and optional blood draw.

Participants will be randomized to one of two arms:

Enhanced Usual Care (EUC), consisting of access to existing usual primary care services such as social determinants of health screenings, referrals to food pantries, and assistance enrolling in food assistance programs. They will be enrolled in a 5-week Hypertension Self-Management Education and Support (SMES) class, which is an existing CDC-endorsed program offered at Eskenazi to provide information and skills for managing hypertension (HTN).

Food Delivery and Cooking PLUS Aerobic Training (FoRKS+), consisting of the same services as EUC plus home-delivered MIND diet ingredient kits and virtual cooking classes for an additional 11 weeks with embedded lessons in kitchen organization, tool use, nutrition, budgeting, and shopping; PLUS aerobic training for an additional 12 weeks of moderate-intensity exercise.

Assessments will be completed at mid-intervention around Week 16, Week 28 as the primary endpoint, and around Week 52 for maintenance evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English
2. Marion County resident
3. 35-75 years
4. Self-identified non-Hispanic and Black/African-American/biracial including African-American
5. Systolic BP of ≥140 in prior 12 months from a primary care visit
6. Ability to see and read street signs (self report)
7. Stable housing with independent access to kitchen, including functional stove or hotplate, oven, refrigerator, and freezer (self report)
8. Activity independence per functional activities questionnaire (FAQ; <3 responses of "Require Assistance" and 0 responses of "Dependent")
9. Normal cognition per six-item screener (SIS; score of ≥ 5)
10. Less than 20min on usual day of moderate or vigorous physical activity
11. Able to exercise safely per abbreviated Exercise Assessment for You (EASY) or primary care provider clearance
12. Mean systolic BP of ≥130 from 3 standard BP measurements taken by research staff following standardized wait periods.

Exclusion Criteria:

1. lives in nursing home
2. diagnosis of dementia or Alzheimer disease or mild cognitive impairment; Parkinson disease; brain tumor/infection/surgery (within the last 10 years with residual symptoms and/or functional loss/deficit, such as impaired learning, memory, or communication); cancer with short life expectancy, or current chemotherapy or radiation therapy; psychosis, schizophrenia, or bipolar disorder
3. ICD 10 code I11/hypertensive heart disease, ICD 10 code I12/hypertensive CKD, ICD 10 code I13/hypertensive heart disease and CKD, ICD 10 code I15, or ICD 10 code I16
4. current or past prescription of donepezil, memantine, rivastigmine, or galantamine
5. alcohol consumption ≥ 8 drinks per week for women, or ≥15 drinks per week for men
6. drug use/abuse (excluding marijuana) per EMR
7. moving out of area during study timeline
8. scheduling conflicts with intervention schedule
9. unwilling to use a touchscreen
10. unwilling to be on video conferencing
11. low communicative ability, functional status, or other disorders (examiner rated) that would interfere with interventions and assessments
12. unable to provide informed consent
13. participation in any lifestyle modification/weight loss program (e.g., Weight Watchers, etc.)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function composite score as measured by individually-administered tests of psychomotor speed, complex sequencing, semantic fluency, interference and list learning and delayed recall at Week 28. | Week 28 post intervention start date
  The cognitive composite is derived from WAIS-IV Symbol Search & Coding, Trail Making Test Part B, Animals-Vegetables-Clothing Naming, Stroop Color-Word, and RBANS Update List Learning and List Recall. The composite will be formed by standardizing each test raw score to the sample baseline mean and standard deviation and then taking an average of the resultant z-scores. These measures will be combined into a single, overall cognitive composite score.
Cognitive function composite score as measured by individually-administered tests of psychomotor speed, complex sequencing, semantic fluency, interference and list learning and delayed recall at Week 52. | Week 52 post intervention start date
  The cognitive composite is derived from WAIS-IV Symbol Search & Coding, Trail Making Test Part B, Animals-Vegetables-Clothing Naming, Stroop Color-Word, and RBANS Update List Learning and List Recall. The composite will be formed by standardizing each test raw score to the sample baseline mean and standard deviation and then taking an average of the resultant z-scores. These measures will be combined into a single, overall cognitive composite score.

SECONDARY OUTCOMES:
Average participant self-ratings of intervention acceptability. | From date of randomization until the date of the final training session or the end of the 28-week intervention, whichever came first.
  Average of individual Likert self-ratings of the interventions (where 1 = very unenjoyable, 2 = not enjoyable, 3 = neutral, 4 = enjoyable, and 5 = very enjoyable) throughout the 28-week intervention.
Participant adherence to treatment. | From date of randomization until the date of the final training session or the end of the 28-week intervention, whichever came first.
  Number of training sessions attended divided by the the total number of sessions available.
Participant adherence to outcome assessments. | End of follow-up at 52-weeks.
  Number of participants completing the outcome assessments divided by the total number randomized.
Number of participants with study-related adverse events (AE) by treatment arm. | From enrollment through end of follow-up at 52-weeks.
  Adverse event count for each study arm

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O Clark, PhD, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No